CLINICAL TRIAL: NCT07139626
Title: Screening and Validation of Serum Biomarkers (SLPI, Serpin E1, CXCL10, CXCL13, Properdin) for Predicting Cardiorenal Syndrome in Patients With Chronic Heart Failure: A Prospective Cohort Study
Brief Title: Screening of Predictive Biomarkers for Cardiorenal Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Haiyan Pan (Other)
Responsible Party: Sponsor-Investigator, Haiyan Pan, Professor and Chief Physician, Department of Cardiology, Affiliated Hospital of Nantong University
Organization: Affiliated Hospital of Nantong University (Other)
Other Study IDs: 2025-K124-01-A
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Cardiorenal Syndrome (CRS)
MeSH Terms: conditions — Cardio-Renal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The specific types of samples to be retained are venous serum samples from all study participants, which are the core specimens for biomarker detection and follow-up analysis. Detailed specifications are as follows:
  1. Source and Collection Volume: Derived from 5-8 mL of venous blood collected from each participant (using serum separation tubes without anticoagulants).
  2. Correspondence to Study Phases:
     * For the Screening Phase (60 participants in CHF-only and CHF+CRS subgroups): 1 tube of serum sample per participant, collected once at baseline.
     * For the Validation Phase (90 participants): 2 tubes of serum samples per participant, collected separately at baseline and 1-year follow-up.
  3. Key Feature for Retention: All retained serum samples are processed to exclude blood cells and clotting factors (via centrifugation at 3000 rpm for 10 minutes at 4°C within 1 hour of collection), ensuring they are suitable for subsequent detection of target biomarkers (SLPI, Serpin E1, CXCL10, CXC

GROUPS / COHORTS (3):
- Screening Phase：Screening CHF-only Subgroup: 30 patients with stable CHF (10 HFrEF, 10 HFmrEF, 10HFpEF) and preserved kidney function (eGFR ≥90mL/min/1.73m' and normal serum creatinine).
  Interventions: Other: This is an observational Study.
- Screening Phase：Screening CHF +CRS Subgroup: 30 patients with stable CHF (10 HFrEF, 10 HFmrEF, 10HFpEF) and established kidney function (eGFR <90mL/min/1.73m' and normal serum creatinine).
  Interventions: Other: This is an observational Study.
- Validation Phase: Validation Cohort (Baseline Normal Renal Function): 90 patients with stable CHF (30 HFrEF, 30 HFmrEF, 30HFpEF) and preserved kidney function (eGFR ≥ 90mL/min/1.73m' and normal serum creatinine) at enrollment. They will be followed for 1 year and reclassified into: Validation CHF-only Subgroup: Remaining with normal renal function after 1 year.
  Validation CRS Subgroup: Developed kidney dysfunction(eGFR <90 mL/min/1.73m' or elevated serum creatinine) after 1 year.
  Interventions: Other: This is an observational Study.

INTERVENTIONS:
Other: This is an observational Study. — This is an observational study with no study-assigned interventions.Only observational measurements (blood collection for biomarker analysis) will be performed without modifying existing treatments.

SUMMARY:
This study aims to explore the predictive value of specific biomarkers for cardiorenal syndrome (CRS) in patients with chronic heart failure (CHF).

Building on previous research using Luminex technology, which identified that serum levels of SLPI, serpin E1, CXCL10, and CXCL13 were significantly higher, while properdin levels were lower in patients with post-cardiac surgery acute kidney injury (AKI) compared to those without renal impairment, this study will further investigate these biomarkers in the context of CRS.

Adults aged 18-75 with stable CHF (including HFrEF, HFmrEF, and HFpEF subtypes) will be conducted in two phases:1. Screening phase: Compare serum levels of the above biomarkers between 30 CHF patients without kidney dysfunction and 30 CHF patients with CRS to identify biomarkers with significant differences. 2. Validation phase: Follow 90 CHF patients with normal kidney function for 1 year, and divide them into CHF-only and CRS groups based on renal function (creatinine and eGFR) after 1 year. The study will verify the predictive value of the screened biomarkers by comparing their levels before and after follow-up, analyzing correlations with NT-proBNP, creatinine, and eGFR, and using receiver operating characteristic (ROC) curves and area under the curve (AUC) to evaluate their predictive efficacy for CRS. The optimal predictive biomarker for this syndrome will be determined.

The participants will:

Provide blood samples for the detection of biomarkers and liver and kidney function indicators.

Receive one year of standardized heart failure treatment. Undergo regular follow-up visits.

DETAILED DESCRIPTION:
This study is a prospective observational cohort study designed to screen and validate the predictive value of five serum biomarkers (secretory leukocyte protease inhibitor [SLPI], Serpin E1, C-X-C motif chemokine ligand 10 [CXCL10], C-X-C motif chemokine ligand 13 [CXCL13], and Properdin) for cardiorenal syndrome (CRS) in patients with stable chronic heart failure (CHF). It builds on prior preclinical and clinical evidence from Luminex technology-based analyses, which identified differential expression of these biomarkers in patients with post-cardiac surgery acute kidney injury (AKI)-suggesting their potential role in mediating cardiorenal crosstalk, a key pathophysiological feature of CRS.

The five target biomarkers are selected based on their mechanistic relevance to CRS pathogenesis:SLPI & Serpin E1: Both are serine protease inhibitors involved in regulating inflammation and endothelial barrier function. Dysregulation of these molecules has been linked to increased renal tubular injury and cardiac interstitial fibrosis-two core processes driving CRS development in CHF. CXCL10 & CXCL13: These chemokines mediate immune cell recruitment (e.g., T cells, B cells) to sites of cardiac and renal injury. Elevated levels in CHF patients may indicate persistent systemic inflammation, a known trigger for progressive cardiorenal dysfunction.Properdin: As a positive regulator of the alternative complement pathway, Properdin contributes to complement system activation. Reduced Properdin levels (observed in post-cardiac surgery AKI) may reflect impaired complement-mediated tissue repair, increasing susceptibility to renal injury in CHF. This panel addresses a critical gap in current CRS research: existing predictive markers (e.g., NT-proBNP, serum creatinine) lack specificity for cardiorenal crosstalk, while these five biomarkers target pathways uniquely involved in the bidirectional damage between the heart and kidneys.

The study is implemented in two sequential phases, with standardized technical protocols to ensure data reliability:1. Screening Phase (Biomarker Differentiation): this phase focuses on identifying biomarkers with significant expression differences between CHF patients with and without CRS. For serum sample processing: Venous blood samples (5 mL) are collected from participants after an 8-hour fasting period, centrifuged at 3,000 rpm for 10 minutes at 4°C to separate serum, and stored at -80°C within 1 hour of collection to avoid biomarker degradation. Biomarker detection uses a multiplex Luminex xMAP assay (custom panel targeting SLPI, Serpin E1, CXCL10, CXCL13, Properdin) with a lower limit of detection (LLOD) ≤ 0.1 pg/mL for each analyte. Assays are run in duplicate, with inter-assay and intra-assay coefficients of variation (CV) controlled at < 10% to ensure reproducibility.

2. Validation Phase (Predictive Efficacy Assessment): this phase validates the predictive performance of screened biomarkers in CHF patients with baseline normal renal function. Key technical procedures include: Longitudinal Sample Tracking: Participants provide serum samples at baseline (enrollment) and 1-year follow-up. Samples are labeled with unique identifiers linked to electronic case report forms (eCRFs) to track renal function (creatinine, eGFR) and biomarker levels over time.

Statistical Validation Framework: Predictive efficacy is evaluated using receiver operating characteristic (ROC) curve analysis, with area under the curve (AUC) calculated to quantify discriminative ability. Biomarker cut-off values for CRS prediction are determined via the Youden index (maximizing sensitivity + specificity). Additionally, Pearson or Spearman correlation analyses are used to assess associations between biomarker levels and clinical indicators (NT-proBNP, creatinine, eGFR), with adjustments for potential confounders (e.g., age, CHF subtype, comorbidities) using multivariable linear regression models.

To account for heterogeneity in CHF pathophysiology, the study stratifies participants by CHF subtype (HFrEF: LVEF ≤ 40%; HFmrEF: LVEF 41-49%; HFpEF: LVEF ≥ 50%) in both phases. This stratification is critical for two technical reasons:1. Biomarker expression may vary by cardiac contractile function (e.g., HFpEF is characterized by myocardial stiffness rather than systolic dysfunction, which may alter inflammatory and complement pathway activation).2. Stratified analyses allow for the evaluation of subtype-specific predictive efficacy-ensuring the identified biomarkers are applicable across the full spectrum of CHF, rather than limited to a single subtype.

All LVEF measurements are standardized using transthoracic echocardiography (TTE) per the 2024 Chinese Heart Failure Diagnosis and Treatment Guidelines, with measurements performed by two independent cardiologists (blinded to biomarker results) to reduce inter-observer variability.

This protocol's technical design prioritizes reproducibility, mechanistic relevance, and clinical applicability-ensuring the validated biomarkers can ultimately be translated into clinical tools for early CRS detection in CHF patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 75 years.
* Diagnosed with stable chronic heart failure (HF) according to the 2024 Chinese Heart Failure Diagnosis and Treatment Guideline.
* HF subtypes include:

HFrEF (LVEF ≤40%), HFmrEF (LVEF 41 - 49%), HFpEF (LVEF ≥50%).

* Willing to provide blood samples for biomarker analysis.
* Able to comply with follow - up visits and study procedures for 12 months.
* Note: For the screening phase, 10 patients will be included for each subtype; for the validation phase, 30 patients will be included for each subtype.

Exclusion Criteria:

* History of long-term dialysis or kidney surgery.
* Acute kidney injury (AKI) within the past 3 months.
* Use of nephrotoxic drugs within the past 3 months.
* Diagnosis of autoimmune diseases (e.g., lupus, rheumatoid arthritis).
* Active malignancy or history of cancer treatment within the past 5 years.
* Acute infectious diseases at the time of enrollment.
* Severe liver dysfunction (e.g., cirrhosis, ALT/AST >3× upper limit of normal).
* Pregnancy or lactation.
* Inability or unwillingness to provide informed consent.
* Participation in another interventional clinical trial within the past 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from chronic heart failure (CHF) patients attending the cardiology outpatient clinics or admitted to the cardiology wards of a tertiary care hospital in China. The study focuses on adults with stable CHF(HFrEF, HFmrEF, HFpEF). The hospital is a regional referral center with a high volume of HF cases, ensuring a diverse and representative sample. Eligible patients will be enrolled based on clinical diagnosis and willingness to participate in biomarker analysis and follow-up assessments.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in serum levels of SLPI, serpin E1, CXCL10, CXCL13, and properdin between the screening CHF - only subgroup and screening CHF + CRS subgroup | At baseline (screening phase).
Predictive efficacy of the screened biomarkers for CRS development in the validation cohort, evaluated by ROC curves and AUC | From enrollment to 1- year follow- up (validation phase).

SECONDARY OUTCOMES:
Correlations between the screened biomarkers and renal function indicators (creatinine, eGFR) | At baseline and 1- year follow- up (validation phase).
Changes in levels of the screened biomarkers between baseline and 1 - year follow - up in the validation CHF - only and validation CRS subgroups | From enrollment to 1- year follow- up (validation phase).
Correlation between serum levels of screened biomarkers and serum NT-proBNP levels in the Validation Phase | At baseline and 1- year follow- up (validation phase).
  Evaluate the correlation between the serum concentration of each screened biomarker (SLPI, Serpin E1, CXCL10, CXCL13, Properdin) and the serum concentration of N-terminal pro-B-type Natriuretic Peptide (NT-proBNP) in participants of the Validation Phase.
  * Measurement Details:
  * Screened biomarkers: Serum concentration (unit: pg/mL), measured by enzyme-linked immunosorbent assay (ELISA) kits (commercially available, validated for sensitivity ≥ 0.1 pg/mL and inter-assay CV < 10%).
  * NT-proBNP: Serum concentration (unit: pg/mL), measured by chemiluminescence immunoassay (CLIA) using an automated clinical chemistry analyzer (e.g., Roche Cobas e601).
  * Correlation Analysis Method: Pearson correlation (for normally distributed data) or Spearman correlation (for non-normally distributed data) will be used to calculate the correlation coefficient (r) and statistical significance (P-value).
Differences in predictive efficacy of the screened biomarkers among CHF subtypes (HFrEF, HFmrEF, HFpEF) | At 1- year follow- up (validation phase).